CLINICAL TRIAL: NCT03368001
Title: Investigating Social Competence in Youth With Autism: A Multisite Randomized Control Trial
Brief Title: Investigating Social Competence in Youth With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Blythe Corbett, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 171153
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SENSE Theatre (Experimental): SENSE Theatre is a peer-mediated, theatre-based intervention targeting social competence in youth with autism spectrum disorder. The 40 hour intervention is comprised of 10 sessions in which trained typically peers are paired with children with autism spectrum disorder (ASD).
  Interventions: Behavioral: SENSE Theatre
- Tackling Teenage Together (Active Comparator): The Tackling Teenage Together is a psychosocial and sexual education program developed for youth with ASD. It is comprised of 10 sessions.
  Interventions: Behavioral: Tackling Teenage Together

INTERVENTIONS:
Behavioral: SENSE Theatre — SENSE Theatre is a peer-mediated, theatre-based intervention targeting social competence in youth with autism spectrum disorder. The 40 hour intervention is comprised of 10 sessions in which trained typically peers are paired with children with autism spectrum disorder (ASD).
  Arms: SENSE Theatre
Behavioral: Tackling Teenage Together — The Tackling Teenage Together is a psychosocial and sexual education program developed for youth with ASD. It is comprised of 10 sessions.
  Arms: Tackling Teenage Together

SUMMARY:
Our treatment, SENSE Theatre, combines several well-documented, effective behavioral strategies and theatre techniques. The proposed project will extend previous findings showing improving improvement in memory for faces. The multisite randomized control trial will include a large sample of 240 children with autism spectrum disorder (ASD) randomly assigned to the experimental (SENSE Theatre) or an active control condition (Tackling Teenage Together).

DETAILED DESCRIPTION:
Recent findings from a randomized control trial (RCT) show immediate between-group effects and evidence of target engagement on the hypothesized mechanism of action, memory for faces, which was evaluated by neuropsychological and event-related potential (ERP) measures. Moreover, the RCT demonstrated treatment effects on social communication skills that generalized to home and community settings. Finally, maintained treatment effects were observed on communication symptoms. The proposed project will extend these findings and provide a stronger test of efficacy using a multisite RCT of SENSE Theatre with a large sample of participants with ASD (8 to 16 years) randomized to an experimental and an active control group. The RCT will assess target engagement of memory for faces and functional change in social interaction with peers. Thus, the overarching aim of the study is to determine whether detected changes in face memory and social interaction are due to the SENSE Theatre treatment and the extent to which these changes generalize and maintain. If predicted results occur, it will provide strong empirical support for a community-based treatment that has generalized effects on a set of core deficits that otherwise have life-long consequences for children and adolescents with ASD.

8/18/2021: Record was updated to delete the outcome measure "Computer memory for faces" as it was not included as a primary outcome variable in the Institutional Review Board (IRB) approved protocol dated 9/13/2017.

ELIGIBILITY:
Inclusion Criteria:

* Children with high-functioning ASD (IQ > or = to 70).

Exclusion Criteria:

* Children who evidence aggression toward other people.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 318 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2023-01-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Alabama, Tuscaloosa, Alabama
  - Stony Brook University, Stony Brook, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Currently sharing with the National Database for Autism Research.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available after study completion and published all primary results.
Access Criteria: Interested investigators must apply to National Database for Autism Research (NDAR) to receive access once it is made available.

REFERENCES:
- [Derived] Corbett BA, White S, Lerner M, Preacher KJ, Klemencic ME, Simmons GL, Pilkington J, Gable P, Gioia A, Key AP. Peers, play, and performance to build social salience in autistic youth: A multisite randomized clinical trial. J Consult Clin Psychol. 2023 Jul;91(7):411-425. doi: 10.1037/ccp0000821. Epub 2023 May 18. PMID 37199977

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Excluded (n = 28) Not meeting inclusion criteria (n = 22) No longer interested (n = 2) Refused to participate (n = 3) Unable to contact (n = 1)
Period: Allocation
Arm/Group | SENSE Theatre | Tackling Teenage Together
Started | 144 | 146
Completed | 120 | 112
Not Completed | 24 | 34
Not completed — Lost to Pretest | 16 | 25
Not completed — Completed Pretest but 0 Intervention sessions | 8 | 9
Period: Posttest
Arm/Group | SENSE Theatre | Tackling Teenage Together
Started | 114 | 93
Completed | 101 | 63
Not Completed | 13 | 30
Not completed — Lost to Posttest | 7 | 11
Not completed — Discontinued Intervention | 6 | 19
Period: Follow-up
Arm/Group | SENSE Theatre | Tackling Teenage Together
Started | 101 | 63
Completed | 95 | 60
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SENSE Theatre | Tackling Teenage Together | Total
Number analyzed (Participants) | 114 | 93 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.62 (1.86) | 12.62 (1.98) | 12.62 (1.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 60
  Male | 83 | 64 | 147
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 15
  Not Hispanic or Latino | 103 | 87 | 190
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 9 | 20
  White | 89 | 74 | 163
  More than one race | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 114 | 93 | 207
Wechsler Abbreviated Scale of Intelligence (WASI) II Full Scale Intelligence Quotient (IQ) [Mean (Standard Deviation); unit: units on a scale] — The Wechsler Abbreviated Scale of Intelligence second edition (WASI-II) is composed of four subtests: Block Design, Vocabulary, Matrix Reasoning, and Similarities. The Full Scale IQ is derived from a summation of the subtests. The IQ Standard Score range is: 40-160. Higher scores mean better outcomes.
  units on a scale | 99.32 (19.25) | 97.28 (17.99) | 98.40 (18.68)
Autism Diagnostic Observation Schedule (ADOS) 2 Severity Scale [Mean (Standard Deviation); unit: units on a scale] — The Autism Diagnostic Observation Schedule, 2nd Edition (ADOS-2) includes a standardized calibrated severity score (CSS). These scores, based on the ADOS-2 total algorithm raw score, range from 1-10, with individuals with ASD ranging from 6-10. The CSS provides a measure of an individual's severity of autistic-like symptoms during when compared to other ASD, regardless of chronological age and language level. Higher scores indicate greater symptom severity.
  units on a scale | 7.25 (1.94) | 7.52 (1.91) | 7.37 (1.92)
IFM Index [Mean (Standard Deviation); unit: µV] — Event-related potential (ERP) Incidental Memory for Faces (IFM) Paradigm is a nonverbal and IQ-independent measure of social information processing. The IFM paradigm targets spontaneous formation of a memory trace for a novel face following repeated presentations. The associated increase in the parietal amplitudes reflects stimulus recall. The unit of measurement is microvolts (µV). IFM index is calculated as the amplitude difference for repeated faces versus single faces, where more positive scores indicate better IFM (greater memory trace for repeated faces).
  µV | -.31 (3.99) | -.17 (3.27) | -0.25 (3.68)
CASS Interested [Mean (Standard Deviation); unit: units on a scale] — The Contextual Assessment of Social Skills (CASS) is an ecologically valid social interaction protocol developed to ascertain several domains of social functioning in youth and young adults with ASD. The CASS features two conditions, Interested (CASS-I) and Bored (CASS-B). Only the CASS-I was used in the study. The DVs analyzed from the CASS included raw scores (range 1-7) for Vocal Expressiveness (varies the tempo, pitch, tone, volume, and/or rhythm of speech), Quality of Rapport (degree of rapport), and Social Anxiety (verbal, nonverbal). Higher scores suggest better functioning.
  units on a scale
    CASS-I Vocal Expressiveness | 4.30 (1.70) | 4.32 (1.56) | 4.31 (1.64)
    CASS-I Quality of Rapport | 4.16 (1.39) | 4.10 (1.21) | 4.13 (1.31)
    CASS-I Social Anxiety | 3.61 (1.61) | 3.99 (1.45) | 3.78 (1.55)
SRS-2 Communication [Mean (Standard Deviation); unit: T-Score] — The Social Responsiveness Scale, Second Edition (SRS-2) is a parent-report measure of behavioral characteristic of autism for ages 2-18 years. Five domain scores are calculated. The standard T-score on the SRS-2 Communication Domain was selected as a treatment outcome. Higher T-scores indicate more impairment.
  The SRS-2 Communication Domain has a mean T-score of 50 with a standard deviation of 10. T-Scores falling in the range of 76 or higher are considered severe, or clinically significant; scores 66-75 are moderate; scores 60-65 are considered mild; and scores 59 or below are average.
  T-Score | 32.33 (8.98) | 32.28 (9.58) | 32.31 (9.23)

OUTCOME MEASURES:

1. Primary Outcome: Developmental Neuropsychological Assessment (NEPSY) Memory for Faces Delayed
Description: A measure of face memory following a delay. Possible score ranges from a scaled score of 1-19 with high scores reflecting better face memory.
Time Frame: Change from baseline to end of treatment (10 weeks).
Population: Unfortunately, collection of the data was not completed and improperly administered at one of the key study sites, rendering the data invalid.
Arm/Group | SENSE Theatre | Tackling Teenage Together
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Incidental Face Memory (IFM) Event-Related Potential (ERP) Task
Description: The IFM involves passive viewing of novel faces one of which repeats. The dependent measure is the difference in ERP amplitude of 250-500 ms time window between the repeated and single face presentation. Positive values indicate better face memory.
Time Frame: Change from baseline to end of treatment (10 weeks) and at two-month follow-up.
Population: Number of participants analyzed at posttest. For follow-up the number of participants was SENSE Theatre N =101 and Tackling Teenage N = 79.
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | SENSE Theatre | Tackling Teenage Together
Number analyzed (Participants) | 107 | 82
µV
  IFM Posttest | .74 (2.39) | -.22 (2.37)
  IFM Follow-up: number analyzed (Participants) | 101 | 79
  IFM Follow-up | .12 (3.05) | .01 (3.27)
Statistical Analysis 1: Comparison: SENSE Theatre vs Tackling Teenage Together; Population models were specified using parameter values derived from past research in tandem with minimal expected effect sizes for the effects of most interest. These models were used to generate 5000 samples for a given N, the models were fit to each sample, and the significance (or not) of key effects was noted. This process was repeated until the target power of at least .80 was reached indicating with 216 participants we would have .82 power; Test type: Other — We used structural equation modeling (SEM), as implemented in Mplus 8.7, as a framework for testing all primary hypotheses. We accounted for any non-independence of observations due to cohort membership by obtaining cluster-robust standard errors using robust maximum likelihood estimation (MLR in Mplus) in tandem with the Type = Complex option available in Mplus, treating cohorts as clusters. All models were structurally saturated, so model fit was necessarily perfect; p = .039, Structural Equation Modeling — IFM Posttest; We used structural equation modeling (SEM), as implemented in Mplus 8.7, as a framework for testing all primary hypotheses
Statistical Analysis 2: Comparison: SENSE Theatre vs Tackling Teenage Together; The indirect effect of SENSE Theatre® vs. TTT through post-test IFM on follow-up Vocal Expressiveness. We adjusted standard errors for cohort, controlled the mediator for individual differences in lag between pretest and posttest for the a path and controlled the outcome for individual differences in lag between pretest to follow-up for the b and c' paths; Test type: Other — The residuals associated with the mediator and outcome were allowed to covary with the lag and pretest scores associated with the outcome, and the residual associated with the outcome was allowed to covary with the lag and pretest scores associated with the mediator; p < 0.05, Structural Equation Model (SEM) — One-tailed significance test; Controlling for Verbal Expressiveness at Pretest and the interval between Pretest and the Followup assessments; Structural Equation Model (SEM) = 0.064, 90% CI 2-sided [0.014 to 0.118] — Estimation parameter represents indirect effect (axb)
Statistical Analysis 3: Comparison: SENSE Theatre vs Tackling Teenage Together; The partially standardized indirect effect of treatment on follow-up Quality of Rapport through posttest Incidental Face Memory. We adjusted standard errors for cohort, controlled the mediator for individual differences in lag (pretest to posttest) and baseline mediator, and controlled the outcome for individual differences in lag (pretest to follow-up) and baseline outcome; Test type: Other — The residual associated with the mediator was allowed to covary with the lag and pretest scores associated with the outcome, and the residual associated with the outcome was allowed to covary with the lag and pretest scores associated with the mediator, yielding a saturated model; p < 0.05, Structural Equation Model (SEM) — One-sided hypothesis test; Controlling for Rapport at Pretest and the interval between Pretest and the Followup assessments; Structural Equation Model (SEM) = 0.032, 90% CI 2-sided [0.002 to 0.087] — Estimation parameter represents indirect effect (axb)
Statistical Analysis 4: Comparison: SENSE Theatre vs Tackling Teenage Together; The partially standardized indirect effect of treatment on follow-up Social Anxiety through posttest IFM. Adjusted standard errors for cohort, controlled the mediator for individual differences in lag between pretest and posttest for the a path and controlled the outcome for individual differences in lag between pretest to follow-up for the b and c' paths; Test type: Other — The residuals associated with the mediator and outcome were allowed to covary with the lag and pretest scores associated with the outcome, and the residual associated with the outcome was allowed to covary with the lag and pretest scores associated with the mediator, yielding a saturated model; p > 0.05, Structural Equation Model (SEM) — One-sided hypothesis test; Controlling for Social Anxiety at Pretest and the interval between Pretest and the Followup assessments; Structural Equation Model (SEM) = 0.005, 90% CI 2-sided [-0.015 to 0.059] — Estimation parameter represents indirect effect (axb)
Statistical Analysis 5: Comparison: SENSE Theatre vs Tackling Teenage Together; The partially standardized indirect effect of treatment on follow-up SRS Communication. We adjusted standard errors for cohort, controlled the mediator for individual differences in lag between pretest and posttest for the a path and controlled the outcome for individual differences in lag between pretest to follow-up for the b and c' paths; Test type: Other — [test comment as in outcome 2, analysis 4]; p > 0.05, Structural Equation Model (SEM) — One-sided hypothesis test; Controlling for SRS-2 Social Communication at Pretest and the interval between Pretest and the Followup assessments; Structural Equation Model (SEM) = -0.0002, 90% CI 2-sided [-0.054 to 0.061] — Estimation parameter represents indirect effect (axb)

3. Secondary Outcome: Social Responsiveness Scale (SRS) Communication
Description: The SRS is a measure of social competence that is administered by parents pertaining to behaviors characteristic of children with autism. Raw scores on the Social Communication domain range from 0 - 66. Higher scores indicate more impairment. Raw scores were used in the analyses. A decrease in scores from pre- to post-treatment suggests a better outcome.
Time Frame: Baseline, post-treatment (10 weeks), and two-month follow-up.
Population: Number of participants analyzed at posttest. Number of participants analyzed at two-month follow-up SENSE Theatre N = 101, Tackling Teenage N = 79.
Measure: Mean (Standard Deviation); unit: Raw scores.
Arm/Group | SENSE Theatre | Tackling Teenage Together
Number analyzed (Participants) | 107 | 82
Raw scores.
  SRS Communication Posttest | 30.33 (9.32) | 30.22 (9.43)
  SRS Communication Follow-up: number analyzed (Participants) | 101 | 79
  SRS Communication Follow-up | 29.74 (9.23) | 29.82 (9.86)
Statistical Analysis 1: Comparison: SENSE Theatre vs Tackling Teenage Together; Test type: Other; p = .490, Structural Equation Modeling — SRS Communication Posttest; [statistical method as in outcome 2, analysis 1]

4. Secondary Outcome: Adaptive Behavior Scales for Children (ABAS)
Description: The ABAS is a parental rating scale pertaining to various adaptive behaviors in a child, such as social and communication skills. Standard scores for the subscales range from 1 to 19. Higher scores reflect better skills in each domain. The primary variable of interest was the Communication subscale, ranging from 1 to 19 with higher scores reflecting better communication skills.
Time Frame: Baseline, post-treatment (10 weeks), and two-month follow-up.
Population: Number of participants analyzed at posttest. One participant in Tackling Teenage had missing data. The number of participants analyzed at two-month follow-up SENSE Theatre N=99, Tackling Teenage N=78. Two participants in SENSE Theatre and one in Tackling Teenage had missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SENSE Theatre | Tackling Teenage Together
Number analyzed (Participants) | 107 | 81
units on a scale
  ABAS Communication Posttest | 6.50 (2.076) | 6.44 (2.185)
  ABAS Communication Followup: number analyzed (Participants) | 99 | 78
  ABAS Communication Followup | 7.32 (5.421) | 6.82 (1.959)
Statistical Analysis 1: Comparison: SENSE Theatre vs Tackling Teenage Together; Test type: Other — Posttest ANCOVA controlling for pre-test scores; p = 0.704, ANCOVA
Statistical Analysis 2: Comparison: SENSE Theatre vs Tackling Teenage Together; Test type: Other — Followup ANCOVA controlling for pretest values; p = 0.406, ANCOVA

5. Secondary Outcome: Contextual Assessment of Social Skills (CASS) Interested
Description: The CASS is an observational measure of social interaction skills with two similar age peers. There are two conditions which include an Interested Condition and a Bored Condition. The behaviors will be coded based on raw scores from 1 to 7 with 7 reflecting better ability. Only the Interested Condition was analyzed.
Time Frame: Baseline, post-treatment (10 weeks), and two-month follow-up.
Population: Number of participants analyzed for Posttest. Number of participants analyzed for Follow-up SENSE Theatre N = 101, Tackling Teenage N = 79.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SENSE Theatre | Tackling Teenage Together
Number analyzed (Participants) | 107 | 82
units on a scale
  Vocal Expressiveness Posttest | 4.29 (1.59) | 3.94 (1.76)
  Vocal Expressiveness Follow-up: number analyzed (Participants) | 101 | 79
  Vocal Expressiveness Follow-up | 4.20 (1.53) | 4.05 (1.75)
  Quality of Rapport Posttest | 4.14 (1.39) | 4.23 (1.66)
  Quality of Rapport Follow-up: number analyzed (Participants) | 101 | 79
  Quality of Rapport Follow-up | 4.26 (1.29) | 4.22 (1.49)
  Social Anxiety Posttest | 4.19 (1.53) | 4.03 (1.59)
  Social Anxiety Follow-up: number analyzed (Participants) | 101 | 79
  Social Anxiety Follow-up | 3.90 (1.40) | 3.77 (1.58)
Statistical Analysis 1: Comparison: SENSE Theatre vs Tackling Teenage Together; Vocal Expressiveness Posttest; Test type: Other; p = .217, Structural Equation Modeling; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: SENSE Theatre vs Tackling Teenage Together; Quality of Rapport Posttest; Test type: Other; p = .448, Structural Equation Modeling; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: SENSE Theatre vs Tackling Teenage Together; Social Anxiety Posttest; Test type: Other; p = .150, Structural Equation Modeling; [statistical method as in outcome 2, analysis 1]

6. Secondary Outcome: Child Behavior Checklist (CBCL)
Description: The CBCL is a parent report measure of a variety of symptom domains relevant for children with autism and related neurodevelopment disorders. T scores range from 40 to 100 with a mean of 50 and a deviation of 10. Primary variable of interest was Social Problems. Higher scores indicate more social problems. T scores of 64 or higher are considered clinically significant.
Time Frame: Baseline, post-treatment (10 weeks), and two-month follow-up.
Population: Number of participants analyzed at posttest. One participant in Tackling Teenage and two participants in SENSE Theatre had missing data. The number of participants analyzed at two-month follow-up SENSE Theatre N=98, Tackling Teenage N=78. Three participants in SENSE Theatre and one in Tackling Teenage had missing data.
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | SENSE Theatre | Tackling Teenage Together
Number analyzed (Participants) | 105 | 80
T score
  CBCL Social Problems Posttest | 64.18 (7.644) | 65.41 (8.422)
  CBCL Social Problems Followup: number analyzed (Participants) | 98 | 78
  CBCL Social Problems Followup | 64.14 (8.445) | 64.65 (8.357)
Statistical Analysis 1: Comparison: SENSE Theatre vs Tackling Teenage Together; Test type: Other — Posttest ANCOVA controlling for pre-test values; p = 0.169, ANCOVA
Statistical Analysis 2: Comparison: SENSE Theatre vs Tackling Teenage Together; Test type: Other — Followup ANCOVA controlling for pretest values; p = 0.555, ANCOVA

ADVERSE EVENTS:
Time Frame: Baseline through study completion (on average, approximately 18 weeks).
Arm/Group | SENSE Theatre | Tackling Teenage Together
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/93
Other Adverse Events (participants affected / at risk) | 0/114 | 0/93

LIMITATIONS AND CAVEATS:
There is data loss due to the Coronavirus -19 pandemic, which resulted in reduction in the number of participants who completed the study, data loss of specific primary variables, and differential attrition between the groups. This is reflected in Participant Flow.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT03368001/Prot_001.pdf
  • Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT03368001/SAP_002.pdf
  • Informed Consent Form (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/01/NCT03368001/ICF_003.pdf